CLINICAL TRIAL: NCT07222709
Title: A Phase 1, Double-blind, Placebo-controlled, First-in-human Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of ABBV-1042 in Healthy Subjects
Brief Title: A Study to Assess the Adverse Events and How Oral ABBV-1042 Moves Through the Body of Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: M25-818
Record Dates: First submitted 2025-10-29; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ABBV-1042

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- ABBV-1042 or Placebo-Group 1 (Experimental): Participants will receive an oral dose of ABBV-1042 or placebo on day 1.
  Interventions: Drug: ABBV-1042; Drug: Placebo
- ABBV-1042 or Placebo-Group 2 (Experimental): Participants will receive an oral dose of ABBV-1042 or placebo on day 1.
  Interventions: Drug: ABBV-1042; Drug: Placebo
- ABBV-1042 or Placebo-Group 3 (Experimental): Participants will receive an oral dose of ABBV-1042 or placebo on day 1.
  Interventions: Drug: ABBV-1042; Drug: Placebo
- ABBV-1042 or Placebo-Group 4 (Experimental): Participants will receive an oral dose of ABBV-1042 or placebo on day 1.
  Interventions: Drug: ABBV-1042; Drug: Placebo
- ABBV-1042 or Placebo-Group 5 (Experimental): Participants will receive an oral dose of ABBV-1042 or placebo on day 1.
  Interventions: Drug: ABBV-1042; Drug: Placebo
- ABBV-1042 or Placebo-Group 6 (Experimental): Participants will receive an oral dose of ABBV-1042 or placebo on day 1.
  Interventions: Drug: ABBV-1042; Drug: Placebo

INTERVENTIONS:
Drug: ABBV-1042 — Oral Solution
Drug: Placebo — Oral Solution

SUMMARY:
This study will assess the adverse events, tolerability, and how oral ascending doses of ABBV-1042 moves through the body of healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* BMI is ≥ 18.0 to ≤ 32.0 kg/m2 after rounding to the tenths decimal at Screening. BMI is calculated as weight in kg divided by the square of height measured in meters.
* Body weight ˃ 45 kg at the time of screening and upon initial confinement.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG

Exclusion Criteria:

* History of suicidal ideation within one year prior to study treatment administration and/or history of suicidal behavior or non-suicidal self-injury within two years prior to study treatment administration as evidenced by any "yes" answer to questions on the Columbia-Suicide Severity Rating Scale (C-SSRS) at the screening visit or upon initial confinement.
* Current or past history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, genitourinary, endocrine (including diabetes mellitus, thyroid disorders), malignancy, hematological, immunological, neurological, or psychiatric disease that, , in the opinion of the investigator, could compromise either participant safety or the results of the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events | Up to approximately 32 days
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Number of Participants with Abnormal Change From Baseline in Vital Sign Measurements | Up to approximately 3 days
  Number of participants with abnormal change from baseline in vital sign measurements like systolic and diastolic blood pressure will be assessed.
Change from Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to approximately 3 days
  The C-SSRS is a clinician-rated instrument that reports the severity of both suicidal ideation and behavior, with a higher score denoting more severe suicidal ideation and behavior.
Number of Participants with Abnormal Change in Physical Examinations | Up to approximately 3 days
  Number of participants with abnormal change in physical examinations in areas like cardiovascular, respiratory, and neurological systems will be assessed.
Number of Participants with Change from Baseline in Electrocardiogram (ECG) | Up to approximately 3 days
  12-lead resting ECG will be recorded.
Number of Participants with Abnormal Change in Clinical Laboratory Test Results Like Hematology will be Assessed | Up to approximately 3 days
  Number of participants with abnormal change in clinical laboratory test results like hematology will be assessed.
Maximum Plasma Concentration (Cmax) of ABBV-1042 | Up to approximately 3 days
  Cmax of ABBV-1042
Time to Cmax (Tmax) of ABBV-1042 | Up to approximately 3 days
  Tmax of ABBV-1042
Apparent terminal phase elimination constant (β) of ABBV-1042 | Up to approximately 3 days
  β of ABBV-1042
Terminal Phase Elimination Half-Life (t1/2) of ABBV-1042 | Up to approximately 3 days
  t1/2 of ABBV-1042
Area under the plasma concentration-time curve from time 0 until the last measurable concentration (AUCt) of ABBV-1042 | Up to approximately 3 days
  AUCt of ABBV-1042
Area under the plasma concentration-time curve from time 0 to infinity (AUCinf) of ABBV-1042 | Up to approximately 3 days
  AUCinf of ABBV-1042

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 279405, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-818